CLINICAL TRIAL: NCT05238363
Title: A Single-arm, Open-Label, Multicenter Phase II Clinical Study to Evaluate Efficacy and Safety of HLX07 (Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) in Patients With Locally Advanced or Metastatic Cutaneous Squamous Cell Carcinoma (CSCC)
Brief Title: The Efficacy and Safety of HLX07 in Locally Advanced or Metastatic Cutaneous Squamous Cell Carcinoma (CSCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX07-CSCC201
Record Dates: First submitted 2022-02-07; First posted 2022-02-14 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Cutaneous Squamous Cell Carcinoma
MeSH Terms: interventions — HLX07

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX07 (Experimental): HLX07 1500mg ivgtt Q3W
  Interventions: Drug: HLX07

INTERVENTIONS:
Drug: HLX07 — HLX07 1500mg ivgtt Q3W
  Other Names: Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection

SUMMARY:
Following basal cell carcinoma, Cutaneous Squamous Cell Carcinoma (CSCC) is the most common skin cancer and its incidence remains on a steady rise. The vast majority of CSCC lesions are treated with surgical resection and have a cure rate exceeding 90 percent in early-stage disease. In stark contrast, the 5-year overall survival rate is below 50% for locally advanced patients and less than 10 percent for those with distant metastases. Although the commonly used cisplatin-based combination chemotherapies may achieve an overall response rate of up to 80%, the efficacy is usually not durable. Moreover, the use of chemotherapy is limited due to the many adverse events, especially in elderly patients, who are the largest population of concern for CSCC. The purpose of this study was to assess safety, efficacy in patients with locally advanced or metastatic CSCC given HLX07 (Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF); be willing to follow and be able to complete all study procedures;
2. Aged ≥ 18 years.
3. Histopathologically or cytologically confirmed diagnosis of locally advanced or metastatic Cutaneous Squamous Cell Carcinoma (CSCC).
4. Measurable lesion according to RECIST v1.1 by IRRC.
5. ECOG score 0-1.
6. Expected survival 12 weeks.
7. For fertile female subjects, the pregnancy test must be negative within 7 days before the first dose.

Exclusion Criteria:

1. Prior systemic anti-EGFR monoclonal antibody therapy.
2. A history of other malignancies within three years, except for cured cervical carcinoma in situ, adenocarcinoma in situ of the breast, or tumors that do not require interventional treatment after radical surgery.
3. Participant has any other histologic type of skin cancer, eg, basal cell carcinoma that has not been definitively treated with surgery or radiation, Bowen's disease, MCC, melanoma.
4. Participants with any prior allogeneic solid organ or bone marrow transplantations.
5. Symptomatic brain or meningeal metastases (unless the patient has been on > treatment for 3 months, has no evidence of progress on imaging within 4 weeks prior to initial administration, and tumor-related clinical symptoms are stable).
6. Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage.
7. Active clinical severe infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier), assessed up to 2 years
  Progression-free survival by independent radiological review committee (IRRC) assessment per RECIST v1.1
ORR | up to 2 years
  Objective response rate by IRRC assessment per RECIST v1.1

SECONDARY OUTCOMES:
OS | from the date of first dose unitl the date of death from any cause，assessed up to 2 years
  Overall survival
DOR | from the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier),assessed up to 2 years
  Duration of response

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No